CLINICAL TRIAL: NCT06229171
Title: InTake Care: Development and Validation of an Innovative, Personalized Digital Health Solution for Medication Adherence Support in Cardiovascular Prevention
Acronym: InTakeCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other); Politecnico di Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09M201
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Treatment Adherence and Compliance; Digital Health
Keywords: Personalized Medicine
MeSH Terms: conditions — Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual practice (No Intervention)
- vocal assistant (Experimental)
  Interventions: Other: adherence support system based on a vocal assistant

INTERVENTIONS:
Other: adherence support system based on a vocal assistant — Participants in the intervention group will receive a vocal assistant device and the instructions/support for the activation of the system at their homes. The device will remind the participant, at the times defined during set-up, which therapy should be taken and with what dosage. The participant will have 30 minutes from the first reminder to confirm vocally that the therapy has been taken, which will otherwise be considered as not having been taken.
  Participants in the control group will receive verbal advice from the physician about the need to follow the treatment recommendations and simple indications on possible solutions to maintain adherence, as by the usual practice of the Centre.
  Arms: vocal assistant

SUMMARY:
Inadequate medication adherence (MA) in chronic conditions, including cardiovascular prevention, represents an important risk factor. The use of new IT technologies in this setting is supposed to be useful to improve patients' adherence, but currently available solutions have significant limitations, including lack of personalization and reliance on expensive ad hoc systems.

This interdisciplinary project aims to verify the hypothesis that in patients on chronic antihypertensive treatment MA can be improved through the implementation of a novel digital health solution for MA monitoring and support, based on inexpensive and user-friendly, commercially available technology (voice assistant), connected with web interface for the physician. The intervention will be personalized based on the creation of Personas, intended as multidisciplinary-based representations of different user types. This approach will be tested in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patients
* History of essential hypertension
* Treatment with at least one antihypertensive drug for which dedicated plasma essay is available
* wireless internet connection available at patients' home
* stable clinical conditions
* written informed consent

Exclusion Criteria:

* insufficient technological literacy to manage vocal assistant
* dementia or significant psychiatric disorders
* conditions significantly limiting vocal communication (deafness, significant speech disorders, poor knowledge of Italian language)
* pregnancy or breastfeeding
* active cancer (except basal cell skin carcinoma)
* upper limb amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Adherence (plasma essay - 3m) | after 3 months of randomized intervention
  Percentage of adherent patients based on plasma essay at follow-up visit

SECONDARY OUTCOMES:
adherence (pill count - 3m) | after 3 months of randomized intervention
  percentage of adherent patients based on pill count adherence (AdhVA) at follow-up visit
adherence (voice assistant - 3m) | after 3 months of randomized intervention
  percentage of adherent patients based on voice assistant adherence (AdhVA) at follow-up visit
adherence (questionnaire - 3m) | after 3 months of randomized intervention
  percentage of adherent patients based on MARS-5I (Medication Adherence Report Scale-5 Italian version) at follow-up visit
Adherence (plasma essay - 5m) | after 5 months
  percentage of adherent patients based on plasma essay at final visit
adherence (pill count - 5m) | after 5 months
  percentage of adherent patients based on pill count adherence (AdhVA) at final visit
adherence (voice assistant - 5m) | after 5 months
  percentage of adherent patients based on voice assistant adherence (AdhVA) at final visit
adherence (questionnaire - 5m) | after 5 months
  percentage of adherent patients based on MARS-5I at final visit
24h Systolic Blood Pressure (3m) | after 3 months of randomized intervention
  24-hour systolic blood pressure (ABPM) at follow-up visit
24h Systolic Blood Pressure (5m) | after 5 months
  24-hour systolic blood pressure (ABPM) at final visit

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Bilo, MD, PhD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- San Luca Hospital, Istituto Auxologico Italiano IRCCS, Milan, Italy